CLINICAL TRIAL: NCT00987402
Title: Surgical Site Infections: a Cluster-randomized, Cross-over Study of the Efficacy of Plain Soap and Water Versus Alcohol-based Rubs for Surgical Hand Preparation
Brief Title: Study of the Efficacy of Plain Soap and Water Versus Alcohol-based Rubs for Surgical Hand Preparation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: World Health Organization (Other); AIC Kijabe Hospital (Other)
Responsible Party: Peter M. Nthumba, M.D., Africa Inland Church Kijabe Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KH-PSW-ABHR
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2009-11

CONDITIONS: Postoperative Wound Infection
Keywords: Surgery; hand scrubbing; post-operative infection; surgical site infection; surgical hand preparation; plain soap and water; alcohol-based hand rub; Cost of surgical hand preparation agent; Side effects of use of hand preparation agent
MeSH Terms: conditions — Surgical Wound Infection | interventions — Water; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plain soap and water (Active Comparator): Surgical hand preparation with plain soap and water
  Interventions: Other: Plain soap and water (PSW)
- Alcohol based hand rubs (Active Comparator): Surgical hand preparation with alcohol based alcohol hand rub
  Interventions: Other: Alcohol-based hand rub (ABHR)

INTERVENTIONS:
Other: Plain soap and water (PSW) — Presence or absence of infection
  Other Names: Plain bar soap; WHO recommended alcohol based hand rub formulation II
  Arms: Plain soap and water
Other: Alcohol-based hand rub (ABHR) — Presence or absence of infection
  Arms: Alcohol based hand rubs

SUMMARY:
Surgical site infections (SSI) constitute a significant health-economic and clinical challenge. The investigators conducted a cluster-randomized, cross-over study to compare the efficacy of plain soap and water (PSW), used ubiquitously across sub-Saharan Africa for surgical hand preparation, to alcohol-based hand rub (ABHR), with SSI rates as the main outcome measure.

A total of 3317 patients undergoing clean and clean-contaminated surgery were included in the study and followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing clean or clean-contaminated surgery at AIC Kijabe Hospital

Exclusion Criteria:

* All patients undergoing contaminated, dirty surgeries and those undergoing repeat procedures within 2 weeks after the initial surgical intervention.
* Patients who did not consent to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3317 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Nthumba, MD, Principal Investigator — AIC Kijabe Hospital
Locations (1):
- Africa Inland Church Kijabe Hospital, Kijabe, Central, Kenya

REFERENCES:
- [Derived] Wood JH, Nthumba PM, Stepita-Poenaru E, Poenaru D. Pediatric surgical site infection in the developing world: a Kenyan experience. Pediatr Surg Int. 2012 May;28(5):523-7. doi: 10.1007/s00383-012-3058-x. PMID 22297835
- [Derived] Nthumba PM, Stepita-Poenaru E, Poenaru D, Bird P, Allegranzi B, Pittet D, Harbarth S. Cluster-randomized, crossover trial of the efficacy of plain soap and water versus alcohol-based rub for surgical hand preparation in a rural hospital in Kenya. Br J Surg. 2010 Nov;97(11):1621-8. doi: 10.1002/bjs.7213. PMID 20878941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing surgery at AIC Kijabe Hospital recruited between January 2007 to November 2007
Pre-assignment Details: Patients who declined consent for participation were excluded, as were those undergoing a second procedure within 2 weeks of the first.
Period: Overall Study
Arm/Group | Plain Soap and Water | Alcohol Based Hand Rubs
Started | 1682 (January 2007, with crossover every 2 months) | 1635 (January 2007 with crossover every 2 months)
Completed | 1596 (86 patients did not have some data, and could not be evaluated) | 1537 (98 patients did not have sufficient data)
Not Completed | 86 | 98
Not completed — Insufficient data entry | 86 | 98

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plain Soap and Water | Alcohol Based Hand Rubs | Total
Number analyzed (Participants) | 1682 | 1635 | 3317
Age Continuous [Mean (Standard Deviation); unit: Participants] | 28 (23) | 29 (19) | 29 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 964 | 908 | 1872
  Male | 718 | 727 | 1445
Region of Enrollment [Number; unit: participants]
  Kenya | 1682 | 1635 | 3317

OUTCOME MEASURES:

1. Secondary Outcome: Cost of Hand Preparation Agent
Description: Average weekly costs were estimated for the plain soap and water used each week in the operating room as well as for the procurement, preparation and dispensing of the alcohol-based handrub to enable a comparison between the two study arms.
Time Frame: 30 days
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Euros

2. Primary Outcome: Surgical Site Infection
Description: 255 (8.1%) patients developed SSIs. Rates for the two study arms were similar (8.3% for alcohol-based handrub versus 8.0% for plain soap and water; odds ratio, 1.03; 95% CI, 0.80 - 1.33).
Time Frame: 30 days post-operatively
Measure: Number; unit: Participants
Arm/Group | Plain Soap and Water | Alcohol Based Hand Rubs
Number analyzed (Participants) | 1682 | 1635
Participants | 128 | 127
Statistical Analysis 1: Comparison: Plain Soap and Water vs Alcohol Based Hand Rubs; Power calculations assumed a 2-sided alpha error of 0.05 and a power of 80%. We performed power calculations using a statistical model for a cluster-randomized trial with 8, 10 or 12 clusters including 6 operating rooms each, with different levels of reduction (10%, 30%, 50%) in surgical site infection rates in the active intervention period. By reaching a sample size of 3133 patients, the study was powered to detect a 30% reduction effect in SSI rates, from 10% to 7%; Test type: Superiority or Other; p < 0.05, generalized estimating equation

ADVERSE EVENTS:
Arm/Group | Plain Soap and Water | Alcohol Based Hand Rubs
Serious Adverse Events (participants affected / at risk) | 0/1596 | 0/1537
Other Adverse Events (participants affected / at risk) | 0/1596 | 0/1537

LIMITATIONS AND CAVEATS:
Most cases, post-discharge monitoring was not conducted by outpatient clinic visits following a standard protocol, some data was not collected, and routine microbiologic cultures were not obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No